CLINICAL TRIAL: NCT02494349
Title: Clinical Trial to Investigate and Compare the Pharmacokinetic Characteristics and Safety/Tolerability After Single Administration of JLP-1207 and Soifenacin/Tamsulosin in Healthy Male Volunteers.
Brief Title: The PK Study of the JLP-1207 and Solifenacin/Tamsulosin in Healthy Male Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeil Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: JLP-1207-P1-PK
Record Dates: First submitted 2015-07-08; First posted 2015-07-10 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2015-07

CONDITIONS: LUTS(Lower Urinary Tract Symptoms); Benign Prostatic Hyperplasia; Overactive Bladder
Keywords: α1-blockers; antimuscarinic agent
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia; Urinary Bladder, Overactive | interventions — Solifenacin Succinate; Tamsulosin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- JLP-1207 (Experimental): JLP-1207 dosing in the fed state(high fat meal)
  Interventions: Drug: JLP-1207
- Solifenacin 5mg+Tamsulosin 0.2mg (Experimental): Solifenacin 5mg+Tamsulosin 0.2mg in the fed state(high fat meal)
  Interventions: Drug: Solifenacin 5mg+Tamsulosin 0.2mg

INTERVENTIONS:
Drug: JLP-1207 — The subjects will receive JLP-1207 under fed(high fat meal) condition. After washout period, the subjects will receive Solifenacin 5mg and Tamsulosin 0.2mg under fed(high fat meal) condition.
  Arms: JLP-1207
Drug: Solifenacin 5mg+Tamsulosin 0.2mg — The subjects will receive Solifenacin 5mg and Tamsulosin 0.2mg under fed(high fat meal) condition. After washout period, the subjects will receive JLP-1207 under fed(high fat meal) condition.
  Arms: Solifenacin 5mg+Tamsulosin 0.2mg

SUMMARY:
The purpose of this study is to investigate and compare the pharmacokinetic characteristics and safety/tolerability between JLP-1207(Solifenacin/Tamsulosin 5mg/0.2mg)and co-administration of Solifenacin and Tamsulosin between Solifenacin and Tamsulosin in healthy male volunteers.

DETAILED DESCRIPTION:
A randomized, open-label, single dose, two-way crossover study.

ELIGIBILITY:
Inclusion Criteria:

* 19~45 years healthy male
* Body weight is over 55kg, BMI measurement 18.0kg/m^2~ 27.0kg/m^2
* Signed informed consent form from to participate voluntarily and to comply with the trial requirements.
* Researchers determined suitable volunteers through physical examination, laboratory tests

Exclusion Criteria:

* History of clinically significant liver, kidneys, nervous system, immune system, respiratory, endocrine disorders or tumor or blood disorders, cardiovascular diseases, mental disorders (mood disorders, obsessive-compulsive disorder, etc.)
* Sitting SBP>150mmHg or <100mmHg, sitting DBP>100mmHg or <60mmHg, after 3 minutes break
* An impossible one who participants in clinical trial by investigator's decision including laboratory test result or another reason.
* Have a gastrointestinal disease history that can affect drug absorption (Crohn's disease ulcers, etc) or surgery (except simple appendectomy or hernia surgery)
* History of drug abuse
* Positive urine drug screening
* Administrated investigational product in a previous clinical trial within 90 days of the first administration day in this study.
* Donated blood within 60 days prior to the first administration day in this study.

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2015-08; Primary Completion 2015-11 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
AUClast, Cmax | 192 hours

SECONDARY OUTCOMES:
AUCinf | 192 hours
Tmax | 192 hours
t1/2 | 192 hours
CL/F | 192 hours
Vd/f | 192 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kyung-sang Yu, M.D., Ph.D., Principal Investigator — Seoul National University Hospital(SNUH)

IPD SHARING:
Plan to Share IPD: No